CLINICAL TRIAL: NCT05509387
Title: Investigating if a Stronger tDCS Intensity is More Effective for Improving Naming Ability in People Living With Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Alzheimer's Society (Other)
Responsible Party: Principal Investigator, Tyler Roncero, Scientific Associate, Baycrest
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #22-19
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4mA Stimulation (Experimental)
  Interventions: Device: transcranial direct current stimulation and naming training
- 2mA Stimulation (Active Comparator)
  Interventions: Device: transcranial direct current stimulation and naming training
- SHAM (Sham Comparator)
  Interventions: Device: transcranial direct current stimulation and naming training

INTERVENTIONS:
Device: transcranial direct current stimulation and naming training — Participants will receive mild stimulation or no stimulation along with naming training

SUMMARY:
There is currently little symptomatic therapy for Alzheimer's Disease (AD) and nothing effective for individuals with Frontotemporal dementia (FTD). However, neuromodulation with transcranial direct current stimulation (tDCS) has the potential to be a clinically effective therapy for both AD and FTD. The challenge now is to specify the parameters and conditions under which tDCS is most effective to transition from the laboratory to clinical medicine. tDCS studies typically report significant group effects despite the variability demonstrated among participants, with some showing clear, meaningful improvement, while others only show statistical improvement or none at all. These variable results may be related to the conventional stimulation intensity level of 2mA. The investigators predict that administering tDCS at 4.0 mA, a more significant number of participants would show a meaningful response, and those who improve at 2mA may improve even more from 4.0mA due to having a larger electric field produced. The investigators aim to test this hypothesis in people with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate AD
* Score between 18 and 25 on the MoCA
* Score on the Cambridge Naming Task during the pre-assessment

Exclusion Criteria:

* No history of stroke or TBI
* No shunts or metal in the body
* No history of significant heart disease, alcoholism and drug use

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Naming Training | 3 months
  The primary outcome measure will be change on the naming lists administered, both a trained version and an untrained version. This change will be measured in terms of the number of images correctly named post-training compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT05509387/Prot_002.pdf
  • Informed Consent Form (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT05509387/ICF_003.pdf